CLINICAL TRIAL: NCT00059605
Title: Phase I Study Of Intravenous DOTAP:Cholesterol-Fus1 Liposome Complex (DOTAP:Chol-fus1) In Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Previously Treated With Chemotherapy
Brief Title: Phase I Study of IV DOTAP: Cholesterol-Fus1 in Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-123
Record Dates: First submitted 2003-04-29; First posted 2003-04-30 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Lung Cancer; NSCLC; SCLC; DOTAP:Chol-fus1; gene; gene transfer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DOTAP:Chol-fus1 (Experimental): Infusion intravenous once every 3 weeks
  Interventions: Genetic: DOTAP:Chol-fus1

INTERVENTIONS:
Genetic: DOTAP:Chol-fus1 — Infusion of DOTAP:Chol-fus1 by vein once every 3 weeks.
  Other Names: DOTAP:Chol-FUS1 Liposomes

SUMMARY:
The goal of this clinical research study is to find out the highest safe dose of DOTAP:Chol-fus1 that can be given to participants in the treatment of non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC). This study is an attempt to transfer a gene (fus1) into cancer cells, using the drug DOTAP:Cholesterol-fus1. Researchers will also study the side effects of this experimental gene transfer at different doses, and will conduct tests to see if there are any effects on tumor size at different doses. Experimental transfer of the fus1 gene into humans has never been tried before.

Objectives:

* Assess the toxicity of DOTAP:Cholesterol-fus1 Liposome Complex (DOTAP:Chol-fus1) administered intravenously.
* To determine the maximal tolerated dose and recommended phase II dose of DOTAP:Chol-fus1 administered intravenously.
* Assess the expression of fus1 following intravenous delivery of DOTAP:Chol-fus1 in tumor and normal bronchial epithelial cell biopsies.
* Assess any anti-cancer activity for DOTAP:Chol-fus1.

DETAILED DESCRIPTION:
DOTAP:Chol-fus1 is a drug that helps transfer the fus1 gene into cancer cells. It is thought that the absence of the fus1 gene may be involved in the development of lung cancer tumors. The idea is to try to replace this gene in lung cancer cells.

Participants in this study must have advanced lung cancer that has worsened after receiving prior chemotherapy. Before treatment begins, participants will have a physical exam. Blood (about 2 tablespoons) and urine tests will be performed. Women able to have children will have a blood pregnancy test. Please note that it is possible that the tumor could cause a "positive" pregnancy test result, when you are not pregnant. If a pregnancy test comes back positive, and for any reason you and/or the research staff believes that this may be an error, additional tests may be done to confirm or rule out pregnancy. The participant's tumor will be measured using CT, PET/CT or MRI scans. Participants will also have an EKG (heart function test) and a MUGA scan or echocardiogram.

A treatment cycle on this study is 3 weeks. Participants will receive pre-medications of dexamethasone and diphenhydramine prior to the infusion of DOTAP:Chol-fus1 to try to lessen the potential reactions to the infusion. The participant will receive a short infusion of DOTAP:Chol-fus1 by vein once every 3 weeks. Participants will be examined by their doctor before each treatment. In addition, participants will return to the clinic on days 2, 3, and 8 after the first dose to have blood tests done, their vital signs checked, and to look for side effects. After every two treatment cycles or 6 weeks, the participant's tumor will be measured using a CT or MRI scan. Participants can continue to receive treatments until the tumor gets worse, side effects become too severe, or a maximum of 6 treatments have been given. Treatment may continue for participants who continue to benefit from the treatment at the end of the planned 6 treatments if the treating physician, the principle investigator, and an advisor from the FDA all agree. Participants will return to the clinic 3 weeks after their last dose of DOTAP:Chol-fus1 to have their vital signs checked and to look for side effects. After all treatments are finished, participants will be contacted every 3 months for an update on their health and to gather information about any other treatment(s) they have received.

Participants entered at a given dose level will not be able to receive a higher dose while on study. A group of 3 participants will receive DOTAP:Chol-fus1 by vein at each dose level. After treating 3 participants at a given dose level, the participants will be observed for 2 weeks to evaluate the toxicity. The information showing if the participants develop severe side effects, referred to as dose-limiting toxicity (DLT), will be recorded for computing the chance of toxicity. This information will be used to help select the dose level for the next group of participants. The goal is to find the dose level where 10% of participants develop severe side effects (dose-limiting toxicity).

All the participants will be treated in a dose-escalation fashion starting from the lowest level. The next dose level can be moved up if calculation of the side effects shows that a higher dose is needed. However, no skipping of doses is allowed.

This is an investigational study. Up to 51 individuals will receive study drug on this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC)
2. For NSCLC subjects: Locally advanced, unresectable, incurable stage IIIB (pleural effusion) or stage IV NSCLC, or recurrent NSCLC that is not potentially curable by radiotherapy or surgery. Patients must have received at least one prior platinum-based chemotherapy regimen for NSCLC. For SCLC subjects: Extensive disease or recurrent disease after initial treatment for limited disease. Patients must have received prior platinum-based chemotherapy or chemoradiotherapy. All subjects: There is no limit to the number of prior chemotherapy regimens received.
3. Preference will be given to patients with tumors amenable to biopsy. In the expansion cohort at MTD, all patients must have tumor amenable to biopsy and must consent to biopsy.
4. Karnofsky Performance Status >= 70%, or Zubrod Performance Status <= 1.
5. Negative serum pregnancy test (serum HCG) if female and of childbearing potential. Since beta-HCG may be falsely elevated as a result of malignancy, women of child-bearing potential who have an elevated serum beta-HCG level are eligible for enrollment if they have two Transvaginal Ultrasound (TVUS) scans one week apart and serial beta-HCG levels two weeks apart that are inconsistent with pregnancy and a Gynecology consult to ensure that the beta- HCG level was at a value high enough to see pregnancy with TVUS. Subjects must agree to practice effective birth control during the study period.
6. Negative serology for Human Immunodeficiency Virus.
7. Patients must be >/= 4 weeks beyond major surgical procedures such as thoracotomy, laparotomy or joint replacement, and must be >/= 1.5 weeks beyond minor surgical procedures such as biopsy of subcutaneous tumors, pleuroscopy, etc, and must not have evidence of wound dehiscence, active wound infection, or comparable major residual complications of the surgery. Absolute neutrophil count (ANC) > 1500 * 10**9/mm**3, platelet count > 100,000 * 10**9/mm**3. Prothrombin time (PT) and Partial thromboplastin time (PTT) < 1.25 times the institutional upper limit of normal.
8. Adequate renal function documented by serum creatinine of <= 1.5 mg/dl or calculated creatinine clearance > 50 ml/min.
9. Adequate hepatic function as documented by serum bilirubin< 1.5 mg/dl and SGOT and SGPT </= 1.5 * upper limit of normal.
10. FEV1 and corrected DLCO of >/= 40% of predicted.
11. Patients with asymptomatic brain metastases that have been treated are eligible if the following criteria are met: No history of seizures in the preceding 6 months. Definitive treatment must have been completed ≥4weeks prior to registration. Subjects must be off steroids that were being administered because of brain metastases or related symptoms for ≥2 weeks. Post-treatment imaging within 2 weeks of registration must demonstrate stability or regression of the brain metastases.
12. Stable cardiac condition with a left ventricular ejection fraction > 50%.
13. Patients must have voluntarily signed an informed consent in accordance with institutional policies.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding.
2. Patients who received investigational therapy, monoclonal antibody such as bevacizumab or cetuximab, or who received radiotherapy to the skull, spine, thorax or pelvis within 30 days of entry into the protocol. Patients are permitted to have received palliative radiotherapy to an extremity provided at least 14 days has elapsed since completion of therapy, provided the patient received no more than 10 radiotherapy fractions and a dose no higher than 30 Gy to that site, and provided skull, spine, thorax or pelvis were not in the radiotherapy field.
3. Patients with brain metastases (except as allowed in inclusion criterion #11). Neurological assessment will be used to determine brain metastases.
4. Active systemic viral, bacterial or fungal infections requiring treatment.
5. Patients with serious concurrent illness or psychological, familial, sociological, geographical, or other concomitant conditions that, in the opinion of the investigator, would not permit adequate follow-up and compliance with the study protocol.
6. Use of any investigational agent within four weeks of study treatment.
7. Prior gene therapy.
8. History of myocardial infarction within 6 months, angina within the past 6 months, or a history of arrhythmias on active therapy.
9. Patients who have received standard chemotherapy with FDA approved agents within 21 days of entry into the protocol.
10. Patients who have received therapy with an oral tyrosine kinase inhibitor (eg, erlotinib) within 14 days prior to entry into the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of DOTAP:Chol-fus1 | Before each dose level (3 weeks); Days 2, 3, and 8 after first dose, blood tests, vital signs, and side effects; and after every two treatment cycles or 6 weeks, tumor measured using CT or MRI scan.

SECONDARY OUTCOMES:
Toxicity of the Intravenous DOTAP:Chol-fus1 complex | Observation for 2 weeks follwing each treatment cycle (3 weeks) for toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: David J. Stewart, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lu C, Stewart DJ, Lee JJ, Ji L, Ramesh R, Jayachandran G, Nunez MI, Wistuba II, Erasmus JJ, Hicks ME, Grimm EA, Reuben JM, Baladandayuthapani V, Templeton NS, McMannis JD, Roth JA. Phase I clinical trial of systemically administered TUSC2(FUS1)-nanoparticles mediating functional gene transfer in humans. PLoS One. 2012;7(4):e34833. doi: 10.1371/journal.pone.0034833. Epub 2012 Apr 25. PMID 22558101
- See also: UT M.D.Anderson Cancer Center — http://www.mdanderson.org